CLINICAL TRIAL: NCT03216304
Title: Drug Interaction Study of Safinamide and a BCRP Substrate, Rosuvastatin, Concomitantly Administered to Healthy Volunteers
Brief Title: Safinamide Steady State Interaction With Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cross Research S.A. (Industry)
Collaborators: Zambon SpA (Industry)
Responsible Party: Principal Investigator, Milko Radicioni, Principal Investigator and Scientific Director, Phase I Unit, Cross Research S.A.
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Z7219J02
Record Dates: First submitted 2017-06-01; First posted 2017-07-13 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-06

CONDITIONS: Healthy
MeSH Terms: interventions — safinamide; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rosuvastatin (Experimental): Film-coated tablets Rosuvastatin will be administered at the dose of 20 mg (single dose at day 1)
  Interventions: Drug: 20 mg rosuvastatin calcium period 1
- safinamide + rosuvastatin (Experimental): Film-coated tablets Safinamide will be administered at the dose 100 mg (once a day for 11 days) Film-coated tablets Rosuvastatin will be administered at the dose of 20 mg (single dose at 12)
  Interventions: Drug: 100 mg safinamide; Drug: 20 mg rosuvastatin calcium period 2

INTERVENTIONS:
Drug: 100 mg safinamide — Safinamide will be administered as follows:
  * Days 5-11: 100 mg safinamide (one Xadago® tablet), once a day
  * Day 12: a single dose of 100 mg safinamide (one Xadago® tablet), immediately followed by a single dose of 20 mg rosuvastatin calcium (one Crestor® tablet)
  * Days 13-15: 100 mg safinamide (one Xadago® tablet) once a day The medication will be orally administered in the morning, at 8:00±1h, under fasting conditions, with 240 mL (total volume) of still mineral water.
  Other Names: Xadago®
  Arms: safinamide + rosuvastatin
Drug: 20 mg rosuvastatin calcium period 1 — Rosuvastatin will be administered as follows:
  - Day 1: a single dose of 20 mg rosuvastatin calcium (one Crestor® tablet)
  Other Names: Crestor®
  Arms: rosuvastatin
Drug: 20 mg rosuvastatin calcium period 2 — - Day 12: a single dose of 20 mg rosuvastatin calcium (one Crestor® tablet) immediately after the safinamide administration
  Other Names: Crestor®
  Arms: safinamide + rosuvastatin

SUMMARY:
To evaluate if safinamide at the steady state, obtained after multiple 100 mg once a day administrations, has an effect on the pharmacokinetics of rosuvastatin, concomitantly administered as a single 20 mg dose, with respect to the pharmacokinetics of 20 mg rosuvastatin administered alone.

DETAILED DESCRIPTION:
Xadago® SmPC reports that safinamide may transiently inhibit BCRP, therefore a time interval of 5 h should be kept between dosing of safinamide and medicinal products that are BCRP substrates with a Tmax ≤ 2 h (e.g. pitavastatin, pravastatin, ciprofloxacin, methotrexate, topotecan, diclofenac or glyburide).

Following a specific request of FDA, the present interaction study in healthy male and female volunteers will be conducted in order to determine if multiple dose administration of safinamide with the BCRP substrate rosuvastatin alters the plasma exposure of rosuvastatin in vivo. Orally administered rosuvastatin, a 3-hydroxy-3-methylglutaryl coenzyme A (HMG-CoA) reductase inhibitor, developed for the treatment of dyslipidaemia, represents a sensitive probe to assess the magnitude of BCRP inhibition. In PK trials in healthy volunteers, rosuvastatin Tmax ranged from 1.7 to 5 h after administration of 10-80 mg doses.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: signed written informed consent before inclusion in the study
2. Sex and age: males and females, 25-55 years old, inclusive
3. Body Mass Index (BMI): 18.5-30 kg/m2, inclusive
4. Vital signs: systolic blood pressure (SBP) 100-139 mmHg, diastolic blood pressure (DBP) 50-89 mmHg, heart rate (HR) 50-90 bpm, measured after 5 min of rest in the sitting position
5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study
6. Contraception and fertility (females only): females of child-bearing potential and with an active sexual life must be using at least one of the following reliable methods of contraception:

   1. A non-hormonal intrauterine device or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit
   2. A male sexual partner who agrees to use a male condom with spermicide
   3. A sterile sexual partner Female participants of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted.

For all female subjects, pregnancy test result must be negative at screening (serum β-HCG test) and day -3 (urine test).

Exclusion Criteria:

1. Contraindications: contraindications to monoamine oxidase-B (MAO-B) inhibitors, antiepileptic drugs, statins and HMG-CoA reductase inhibitors
2. Origin: Asian subjects
3. Electrocardiogram (ECG 12-leads, supine position): clinically significant abnormalities
4. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study; albinism
5. Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness
6. Allergy: ascertained or presumptive hypersensitivity to the active principles and/or formulations' ingredients; hypersensitivity or history of anaphylaxis to drugs or allergic reactions in general, which the investigator considers may affect the outcome of the study. Subjects with rare hereditary problems of galactose intolerance, the Lapp lactose deficiency or glucose-galactose malabsorption
7. Diseases: significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine, neurological or musculoskeletal diseases that may interfere with the aim of the study
8. Medications: medications, including over the counter medications and herbal remedies, for 2 weeks before the start of the study. In particular statins and HMG-CoA reductase inhibitors in the 4 weeks before the screening visit; medicinal products that are BCRP substrates; ciclosporin, protease inhibitors, gemfibrozil and other lipid-lowering products, ezetimibe, antacid containing aluminium and magnesium hydroxide, erythromycin and other medicinal products according to the information reported in rosuvastatin SmPC, in the 4 weeks before the screening visit; treatment with morphine or other similar opioids, whose concomitant use with MAO-B inhibitors is contraindicated, SSRIs, SNRIs, tri- or tetracyclic antidepressant, tramadol, pethidine, dextromethorphan, MAO inhibitors (e.g. selegiline), meperidine derivatives and antiepileptic drugs in the 4 weeks before the screening visit; treatment with any known enzyme inhibiting or inducing agent within 4 weeks preceding the screening visit. Hormonal contraceptives
9. Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study
10. Blood donation: blood donations for 3 months before this study
11. Drug, alcohol, caffeine, tobacco: history of drug, alcohol [>1 drink/day for females and >2 drinks/day for males, defined according to the USDA Dietary Guidelines 2015-2020], caffeine (>5 cups coffee/tea/day) or tobacco abuse (≥10 cigarettes/day)
12. Drug test: positive drug test at screening or day -3
13. Alcohol breath test: positive alcohol breath test at day -3
14. Diet: abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians; intake of alcohol, grapefruit or grapefruit juice, apple or orange juice, vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, brussels sprouts, mustard), and charbroiled meats for 1 week before the start of the study
15. Pregnancy (females only): positive or missing pregnancy test at screening or day -3, pregnant or lactating women

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Transporter-Mediated Interaction (TMI) between safinamide (investigational drug) and rosuvastatin (selected BCRP substrate) defined as ANOVA comparison between AUC of treatments (co-administration / rosuvastatin alone) | 96 hours
  Transporter-Mediated Interaction (TMI) between safinamide (investigational drug) and rosuvastatin (selected BCRP substrate) evaluated after the FDA - CDER Draft Guidance on Drug Interaction Studies of February 2012. Blood samples will be collected at different time points up to 96 h and the concentrations of rosuvastatin will be measured after single administration of a 20 mg dose with and without co-administration of multiple 100 mg doses of safinamide in a cross-over design. The Area Under the Curve (AUC), calculated with a non-compartmental method will be used as metrics for the plasma rosuvastatin extent of exposure. The parametric point estimators (PEs) for the ratios of treatments (co-administration / rosuvastatin alone) and the 90% confidence intervals will be calculated using the adjusted least squares means (LSMEANS) from an Analysis of variance (ANOVA) on rosuvastatin AUC. Presence of a TMI will be defined as an upper limit of the 90% confidence interval above 125.00.

SECONDARY OUTCOMES:
Transporter-Mediated Interaction (TMI) between safinamide (investigational drug) and rosuvastatin (selected BCRP substrate) defined as ANOVA comparison between Cmax of treatments (co-administration / rosuvastatin alone) | 96 hours
  Transporter-Mediated Interaction (TMI) between safinamide (investigational drug) and rosuvastatin (selected BCRP substrate). Blood samples will be collected at different time points up to 96 h and the concentrations of rosuvastatin will be measured after single administration of a 20 mg dose with and without co-administration of multiple 100 mg doses of safinamide in a cross-over design. The Peak Concentration (Cmax), calculated with a non-compartmental method will be used as one of the metrics for the plasma rosuvastatin rate of exposure. Secondary criteria for TMI presence will be the same as for the AUC.
Transporter-Mediated Interaction (TMI) between safinamide (investigational drug) and rosuvastatin (selected BCRP substrate) defined as as non-parametric comparison between Tmax of treatments (co-administration / rosuvastatin alone) | 96 hours
  Transporter-Mediated Interaction (TMI) between safinamide (investigational drug) and rosuvastatin (selected BCRP substrate). Blood samples will be collected at different time points up to 96 h and the concentrations of rosuvastatin will be measured after single administration of a 20 mg dose with and without co-administration of multiple 100 mg doses of safinamide in a cross-over design. The Time to the Peak Concentration (Tmax), calculated with a non-compartmental method will be used as one of the metrics for the plasma rosuvastatin rate of exposure. Secondary criteria for TMI presence interaction will be a significant p-value (i.e. >0.05) obtained from a non-parametric Wilcoxon signed-rank test on the Tmax parameter.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 96 hours
  Treatment emergent adverse events (TEAEs), vital signs (blood pressure and heart rate), body weight, electrocardiogram and laboratory parameters will be considered for safety and tolerability assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, MD, Principal Investigator — CROSS Research SA, Phase I Unit, Via FA Giorgioli 12, 6864 Arzo Switzerland
Locations (1):
- CROSS Research SA, Phase I Unit, Arzo, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: CROSS Research — http://www.croalliance.com/